CLINICAL TRIAL: NCT04082702
Title: Reducing Obesity in African American Women Through Lifestyle Enhancement
Brief Title: Better Me Within Trial to Improve Lifestyle Behaviors in African Americans
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Baylor Research Institute (Other)
Collaborators: University of North Texas Health Science Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: P20MD006882-2; P20MD006882 (NIH)
Record Dates: First submitted 2019-08-29; First posted 2019-09-09 (Actual); Last update posted 2019-12-11 (Actual); Status verified 2019-08

CONDITIONS: Obesity; Pre-diabetes
Keywords: CBPR; DPP; African-American; Women; Obesity; Pre-diabetes
MeSH Terms: conditions — Obesity; Glucose Intolerance

STUDY DESIGN:
Intervention Model Description: This study uses a prospective, 2-group, randomized nested (by church) design with eleven congregations, comparing a healthy weight management program with a pastor/church leader component (Intervention) to a healthy weight management program without a pastor/church component (Control). Focus groups were conducted with a sample of 64 participants for understanding needs, perspectives and barriers to healthy weight management. A total of 221 overweight and obese female participants from about 11 churches (approximately 25-30 individuals per church) were recruited and participated in this study following the protocols. The DPP Curriculum includes an intervention phase (approximately weekly for 4 months) and maintenance phase (once or twice a month for 6 months). Faith components (handouts and mini-sermon) are only used by the treatment (intervention) group through both the intervention and maintenance phase.
Who Masked: Outcomes Assessor
Masking Description: Research personnel involved in delivering interventions were not allowed to facilitate the outcome measures. Project coordinator, key personnel, and trained volunteers (which included graduate students) collected all the data elements. Statisticians and data coordinators were blinded of intervention group assignments of the participants until the end of the study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Faith-enhanced DPP (Experimental): A total of six churches were randomized to this arm that included 119 participants and received 10-month DPP with faith components.
  Interventions: Behavioral: Faith-enhanced diabetes prevention program
- Standard DPP (Active Comparator): A total of five churches were randomized to this arm that included 102 participants who received the standard DPP on the church settings.
  Interventions: Behavioral: Standard diabetes prevention program

INTERVENTIONS:
Behavioral: Faith-enhanced diabetes prevention program — The faith-enhanced curriculum was faith-based and developed using CBPR approaches. The Faith-DPP condition included delivery of the DPP. The group intervention was delivered by one to two trained peers from the church and consisted of 16 weekly group meetings followed by 6 bi-monthly or monthly maintenance sessions. The faith enhanced curriculum included five strategies: 1) a mini sermon (~15 min in length) delivered by a pastor (head pastors were required to deliver at least one per month), first lady, or church leader (pastor associate, deacon, elder, etc.), 2) a memory verse, 3) in class or take-home faith activity (application of faith principles), 4) promises to remember, and 5) scripture and prayer integrated into participant curriculum and facilitator materials. These five faith enhancements were developed by the CAB to enhance the DPP's weekly learning objectives, which resulted in faith components specifically linked to each week of DPP content.
  Arms: Faith-enhanced DPP
Behavioral: Standard diabetes prevention program — The S-DPP condition was faith-placed, a secular program (the DPP) held at an faith-based organization. This condition received the same diabetes prevention program (DPP) as the Faith-DPP, but did not receive any faith enhancements or pastor involvement.
  Arms: Standard DPP

SUMMARY:
This study describes a community-based participatory research (CBPR) approach to design a novel faith-enhancement to the diabetes prevention program (DPP) for AA women. A long-standing CBPR partnership designed the faith-enhancement from focus group data. The faith components were specifically linked to weekly DPP learning objectives to strategically emphasize behavioral skills with religious principles. Using a CBPR approach, the Better Me Within trial was able to enroll 12 churches, screen 333 AA women, and randomize 221 after collection of objective eligibility measures. A prospective, randomized, nested by church, design was used to evaluate the faith-enhanced DPP as compared to a standard DPP on weight, diabetes and cardiovascular risk, over a 16-week intervention and 10-month follow up.

DETAILED DESCRIPTION:
Reducing obesity positively impacts diabetes and cardiovascular risk; however, evidence-based lifestyle programs, such as the diabetes prevention program (DPP), show reduced effectiveness in African American (AA) women. In addition to an attenuated response to lifestyle programs, AA women also demonstrate high rates of obesity, diabetes, and cardiovascular disease. To address these disparities, enhancements to evidence-based lifestyle programs for AA women need to be developed and evaluated with culturally relevant and rigorous study designs. This study describes a community-based participatory research (CBPR) approach to design a novel faith-enhancement to the DPP for AA women. A long-standing CBPR partnership designed the faith-enhancement from focus group data (N=64 AA adults) integrating five components: a brief pastor led sermon, memory verse, in class or take-home faith activity, promises to remember, and scripture and prayer integrated into participant curriculum and facilitator materials. The faith components were specifically linked to weekly DPP learning objectives to strategically emphasize behavioral skills with religious principles. Using a CBPR approach, the Better Me Within trial was able to enroll 12 churches, screen 333 AA women, and randomize 221 (Mean age =48.8 ±11.2; Mean BMI =36.7 ±8.4; 52% technical or high school) after collection of objective eligibility measures. A prospective, randomized, nested by church, design was used to evaluate the faith-enhanced DPP as compared to a standard DPP on weight, diabetes and cardiovascular risk, over a 16-week intervention and 10-month follow up. This study provides essential data to guide enhancements to evidence-based lifestyle programs for AA women who are at high risk for chronic disease.

ELIGIBILITY:
Inclusion Criteria:

* Identify as African-American
* Female
* 18 years of age or older
* Parishioner at enrolled church
* Overweight or obese
* Willingness to participate in a 10-month study.

Exclusion Criteria:

* Currently attending a weight loss program
* Diagnosed with diabetes
* Medical condition that interfered with physical activity or dietary changes
* Plans to move in the next 10 months.

Ages: 18 Years to 120 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Only female participants were eligible to enroll in this study due to their higher risk for obesity and diabetes.
Enrollment: 221 (Actual)
Dates: Start 2013-02-22 (Actual); Primary Completion 2017-05-01 (Actual); Study Completion 2017-05-31 (Actual)

PRIMARY OUTCOMES:
Body weight | Baseline
  Weight (lbs) was collected with a digital scale in light clothing with shoes removed. Weight was collected twice and the average was computed. Height was also measured using the same protocol to calculate the BMI (body-mass index).
Body weight | 4-month
  Weight (lbs) was collected with a digital scale in light clothing with shoes removed. Weight was collected twice and the average was computed. Height was also measured using the same protocol to calculate the BMI (body-mass index).
Body weight | 10-month
  Weight (lbs) was collected with a digital scale in light clothing with shoes removed. Weight was collected twice and the average was computed. Height was also measured using the same protocol to calculate the BMI (body-mass index).
Waist circumference: Number of participants above the recommended level | Baseline
  Waist circumference was taken at the top of the pelvis (e.g., above the uppermost lateral border of the right ilium) with a measuring tape twice and averaged.
Waist circumference: Number of participants above the recommended level | 4-month
  Waist circumference was taken at the top of the pelvis (e.g., above the uppermost lateral border of the right ilium) with a measuring tape twice and averaged.
Waist circumference: Number of participants above the recommended level | 10-month
  Waist circumference was taken at the top of the pelvis (e.g., above the uppermost lateral border of the right ilium) with a measuring tape twice and averaged.

SECONDARY OUTCOMES:
Fasting glucose | Baseline
  Fasting glucose was measured with the Cholestech LDX system
Fasting glucose | 4-month
  Fasting glucose was measured with the Cholestech LDX system
Glycated Hemoglobin A1c | Baseline
  Glycated hemoglobin A1C was measured with Bayer A1c Now + Multi-Test A1c System.
Glycated Hemoglobin A1c | 4-month
  Glycated hemoglobin A1C was measured with Bayer A1c Now + Multi-Test A1c System.
Low-density lipoprotein cholesterol (LDL) | Baseline
  LDL was measured with a fasting blood sample obtained by finger stick with the Cholestech LDX system
Low-density lipoprotein cholesterol (LDL) | 4-month
  LDL was measured with a fasting blood sample obtained by finger stick with the Cholestech LDX system
High-density lipoprotein cholesterol (HDL) | Baseline
  HDL was measured with a fasting blood sample obtained by finger stick with the Cholestech LDX system.
High-density lipoprotein cholesterol (HDL) | 4-month
  HDL was measured with a fasting blood sample obtained by finger stick with the Cholestech LDX system.
Blood pressure | Baseline
  Blood pressure was collected with an automated blood pressure device following a seated 5 min rest in a quiet area. Two measurements were taken following Eighth Joint National Committee protocols and averaged.
Blood pressure | 4-month
  Blood pressure was collected with an automated blood pressure device following a seated 5 min rest in a quiet area. Two measurements were taken following Eighth Joint National Committee protocols and averaged.
Blood pressure | 10-month
  Blood pressure was collected with an automated blood pressure device following a seated 5 min rest in a quiet area. Two measurements were taken following Eighth Joint National Committee protocols and averaged.
Dietary patterns: Total energy (Kcal), total fat (gram), total sodium (milligram) intake on a typical day | Baseline
  Diet was measured with the Lower Mississippi Delta Nutrition Intervention Research Initiative (Delta NIRI) food frequency questionnaire. Data is scanned and analyzed by Northeastern University's Dietary Assessment Center. Total energy, fat, sodium, and other dietary components were estimated from the questionnaire.
  Desired total energy (Kcal) (range: 500 to 10,000) intake is defined as 2000 Kcal or less.
  Desired fat (gram) (range: 10 to 500) intake is defined as 77 gram or less. Desired sodium (milligram) (range: 100 to 20,000) intake is defined as 2300 milligram or less.
Dietary patterns: Total energy (Kcal), total fat (gram), total sodium (milligram) intake on a typical day | 4-month
  Diet was measured with the Lower Mississippi Delta Nutrition Intervention Research Initiative (Delta NIRI) food frequency questionnaire. Data is scanned and analyzed by Northeastern University's Dietary Assessment Center. Total energy, fat, sodium, and other dietary components were estimated from the questionnaire.
  Desired total energy (Kcal) (range: 500 to 10,000) intake is defined as 2000 Kcal or less.
  Desired fat (gram) (range: 10 to 500) intake is defined as 77 gram or less. Desired sodium (milligram) (range: 100 to 20,000) intake is defined as 2300 milligram or less.
Physical activity: Total number of active minutes per week | Baseline
  Physical activity was measured by self-report with the Past Week Modifiable Physical Activity Questionnaire. A total of all physical activity minutes was calculated from the questionnaire.
  Desired level of physical activity is defined as 150 minutes or more per week.
Physical activity: Total number of active minutes per week | 4-month
  Physical activity was measured by self-report with the Past Week Modifiable Physical Activity Questionnaire. A total of all physical activity minutes was calculated from the questionnaire.
  Desired level of physical activity is defined as 150 minutes or more per week.
Physical activity | 10-month
  Physical activity was measured by self-report with the Past Week Modifiable Physical Activity Questionnaire. A total of all physical activity minutes was calculated from the questionnaire.
  Desired level of physical activity is defined as 150 minutes or more per week.
Estradiol (pg/mL) | Baseline
  Saliva collected in 4 consecutive weeks and sent to a laboratory to assay
Estradiol (pg/mL) | 4-month
  Saliva collected in 4 consecutive weeks and sent to a laboratory to assay
Cortisol (ng/mL) | Baseline
  Fasting morning saliva sent to a laboratory to assay
Cortisol (ng/mL) | 4-month
  Fasting morning saliva sent to a laboratory to assay

CONTACTS AND LOCATIONS:
Overall Officials: Heather Kitzman, PhD, Principal Investigator — Baylor Scott and White Health
Locations (1):
- UNT Health Science Center, Fort Worth, Texas, United States

IPD SHARING:
Plan to Share IPD: Yes
Contact site contact person
Supporting Information: Study Protocol, SAP, ICF

REFERENCES:
- [Background] Kitzman H, Dodgen L, Mamun A, Slater JL, King G, Slater D, King A, Mandapati S, DeHaven M. Community-based participatory research to design a faith-enhanced diabetes prevention program: The Better Me Within randomized trial. Contemp Clin Trials. 2017 Nov;62:77-90. doi: 10.1016/j.cct.2017.08.003. Epub 2017 Aug 12. PMID 28807739
- [Background] Tan M, Mamun A, Kitzman H, Mandapati SR, Dodgen L. Neighborhood Disadvantage and Allostatic Load in African American Women at Risk for Obesity-Related Diseases. Prev Chronic Dis. 2017 Nov 22;14:E119. doi: 10.5888/pcd14.170143. PMID 29166248
- [Derived] Kitzman H, Mamun A, Dodgen L, Slater D, King G, King A, Slater JL, DeHaven M. Better Me Within Randomized Trial: Faith-Based Diabetes Prevention Program for Weight Loss in African American Women. Am J Health Promot. 2021 Feb;35(2):202-213. doi: 10.1177/0890117120958545. Epub 2020 Sep 18. PMID 32945175
- [Derived] Mamun A, Kitzman H, Dodgen L. Reducing metabolic syndrome through a community-based lifestyle intervention in African American women. Nutr Metab Cardiovasc Dis. 2020 Sep 24;30(10):1785-1794. doi: 10.1016/j.numecd.2020.06.005. Epub 2020 Jun 12. PMID 32605881